CLINICAL TRIAL: NCT00559988
Title: The IMPACT of BIOTRONIK Home Monitoring Guided Anticoagulation on Stroke Risk in Patients With ICD and CRT-D Devices
Brief Title: Combined Use of BIOTRONIK Home Monitoring and Predefined Anticoagulation to Reduce Stroke Risk
Acronym: IMPACT
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Biotronik, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IMPACT
Record Dates: First submitted 2007-11-15; First posted 2007-11-19 (Estimated); Results first posted 2014-06-23 (Estimated); Last update posted 2017-12-05 (Actual); Status verified 2017-11

CONDITIONS: Atrial Fibrillation; Atrial Flutter; Stroke; Embolism, Systemic Arterial; Major Bleeding
Keywords: Implanted Cardioverter Defibrillator; Cardiac Resynchronization Therapy Defibrillator; Home Monitoring; Oral Anticoagulation
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter; Stroke; Embolism

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Home Monitoring Guided OAC (Experimental): Home Monitoring is fully enabled and continuous remote surveillance data is available to investigators. Patients will be treated according to a predefined anticoagulation plan, which uses the total duration of AF/AFL combined with patients' CHADS2 score to determine the start, stop, and restart of OAC.
  Interventions: Drug: Home Monitoring Guided OAC
- Physician-Directed OAC (Active Comparator): In Control (Group 2), Home Monitoring is active for Safety Net alerts, but the remote AF/AFL data is not revealed to the patient or treating physician. These patients receive physician-directed OAC consistent with current standards of care.
  Safety Net data include:
  * ERI/EOS
  * Special Implant Status
  * Implant in Backup Mode (ROM)
  * VT/ VF Detection Inactive
  * Emergency Pacing
  * 250 Ω > RV Pacing Impedance > 1500 Ω
  * Symptomatic VT/VF therapies including both ATP and shock
  * VT/VF storm
  * HM transmission failure >3 days
  Interventions: Drug: Physician-Directed OAC

INTERVENTIONS:
Drug: Home Monitoring Guided OAC — Active monitoring for atrial episodes through the automatic HM notifications (email, fax, short message service) is required. If the total duration over 48 consecutive hours reaches the predefined anticoagulation condition, and AF/AFL diagnosis is confirmed using the IEGM online, the site instructs the patient by telephone to start OAC. Clinicians continue to monitor patients using HM, and if freedom from AF/AFL reaches the predefined interval, stop of OAC therapy is requested over the telephone. Following stop of anticoagulation, any recurrence of AF/AFL requires restart of OAC therapy.
  OAC drugs used: Dabigatran etexilate, Rivaroxaban, Warfarin, other approved VKA
  Arms: Home Monitoring Guided OAC
Drug: Physician-Directed OAC — Patients will receive physician-directed anticoagulation therapy based on conventional criteria.
  OAC drugs used: Dabigatran etexilate, Rivaroxaban, Warfarin, other approved VKA
  Arms: Physician-Directed OAC

SUMMARY:
The IMPACT Study will investigate the potential clinical benefit of the combined use of BIOTRONIK Home Monitoring (HM) technology and a predefined anticoagulation plan compared to conventional device evaluation and physician-directed anticoagulation in patients with implanted dual-chamber defibrillators or cardiac resynchronization therapy devices.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) and atrial flutter (AFL) are common cardiac arrhythmias associated with an increased incidence of stroke in patients with additional risk factors. Oral Anticoagulation (OAC) reduces stroke risk, but because these arrhythmias are frequently intermittent and asymptomatic, start of OAC therapy is often delayed until electrocardiographic documentation is obtained.

Technological advances in implanted dual-chamber cardioverter defibrillator (ICD) or cardiac resynchronization therapy defibrillator (CRT-D) devices allow early detection and real time verification of AF/AFL with intracardiac electrograms (IEGM) automatically transmitted to the clinicians. Such remote diagnostic capability might be particularly relevant in patients with asymptomatic AF by allowing timely treatment. Compared to conventional periodic, (e.g., quarterly) office device evaluation, daily remote monitoring may prove superior for diagnosis of AF and prophylactic treatment of thromboembolism.

The start, stop and restart of OAC based on a predefined atrial rhythm-guided strategy in conjunction with a standard risk-stratification scheme could lead to better clinical outcomes compared with conventional clinical care. The study is designed to demonstrate a risk reduction of both thromboembolism proximate to episodes of documented AF/AFL and bleeding potentiated by chronic OAC in the absence of AF. Verification of this premise would impact the clinical practice, providing evidence to physicians for the use of HM to guide OAC in patients with AF/AFL. The results of this study should demonstrate the clinical value of wireless remote surveillance of the cardiac rhythm and may define the critical threshold of AF/AFL burden warranting OAC or antiarrhythmic drug therapy in patients at risk of stroke

ELIGIBILITY:
Key Inclusion Criteria:

* Candidates for implantation of, or already implanted with, a BIOTRONIK Lumax HF-T or DR-T device
* Documented P wave mean amplitude ≥ 1.0 mV (sinus rhythm) or ≥ 0.5 mV (AF) at enrollment, if previously implanted
* CHADS2 risk score ≥ 1
* Able and willing to follow OAC therapy if the indication develops during the course of the trial
* Able to utilize the HM throughout the study

Key Exclusion Criteria:

* Permanent AF
* History of stroke, transient ischemic attack (TIA) or systemic embolism and documented AF or AFL
* Currently requiring OAC therapy for any indication
* Patients who underwent successful AF ablation (sinus rhythm restored) and have not completed a minimum of 3 months of OAC therapy
* Known, current contraindication to use of eligible OAC
* Long QT or Brugada syndrome as the sole indication for device implantation
* Life expectancy less than the expected term of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2718 (Actual)
Dates: Start 2008-02; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan L Halperin, M.D., Study Chair — Mount Sinai Medical Center, New York, NY; John Ip, M.D., Study Chair — Thoracic & Cardiovascular Healthcare Foundation, Lansing, MI
Locations (80):
- United States (73):
  - Phoenix, Arizona
  - Scottsdale, Arizona
  - Anaheim, California
  - Fremont, California
  - Santa Barbara, California
  - Torrance, California
  - Ventura, California
  - Aurora, Colorado
  - Boulder, Colorado
  - Newark, Delaware
  - Davenport, Florida
  - Daytona Beach, Florida
  - Kissimmee, Florida
  - Melbourne, Florida
  - Sarasota, Florida
  - St. Petersburg, Florida
  - Zephyrhills, Florida
  - Chicago, Illinois
  - Elk Grove Village, Illinois
  - Maywood, Illinois
  - Fort Wayne, Indiana
  - Valparaiso, Indiana
  - Shawnee Mission, Kansas
  - Lexington, Kentucky
  - Louisville, Kentucky
  - Owensboro, Kentucky
  - Hammond, Louisiana
  - Lafayette, Louisiana
  - New Orleans, Louisiana
  - Bangor, Maine
  - Lewiston, Maine
  - Cumberland, Maryland
  - Boston, Massachusetts
  - Burlington, Massachusetts
  - Worcester, Massachusetts
  - Ann Arbor, Michigan
  - Bay City, Michigan
  - Lansing, Michigan
  - Lapeer, Michigan
  - Saginaw, Michigan
  - Ypsilanti, Michigan
  - Minneapolis, Minnesota
  - Tupelo, Mississippi
  - Kansas City, Missouri
  - Osage Beach, Missouri
  - St Louis, Missouri
  - Omaha, Nebraska
  - Ridgewood, New Jersey
  - New York, New York
  - Durham, North Carolina
  - Hickory, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Kettering, Ohio
  - Middletown, Ohio
  - Toledo, Ohio
  - Westlake, Ohio
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Tualatin, Oregon
  - Abington, Pennsylvania
  - Philadelphia, Pennsylvania
  - Phoenixville, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Greenville, South Carolina
  - Rock Hill, South Carolina
  - Cookeville, Tennessee
  - Germantown, Tennessee
  - Nashville, Tennessee
  - Corpus Christi, Texas
  - Houston, Texas
  - Humble, Texas
  - Kingwood, Texas
- Wahroonga, Australia
- Canada (2):
  - Montreal, Quebec
  - Sherbrooke, Quebec
- Aarhus, Denmark
- Germany (2):
  - Tübingen
  - Villingen
- Birmingham, United Kingdom

REFERENCES:
- [Derived] Martin DT, Bersohn MM, Waldo AL, Wathen MS, Choucair WK, Lip GY, Ip J, Holcomb R, Akar JG, Halperin JL; IMPACT Investigators. Randomized trial of atrial arrhythmia monitoring to guide anticoagulation in patients with implanted defibrillator and cardiac resynchronization devices. Eur Heart J. 2015 Jul 7;36(26):1660-8. doi: 10.1093/eurheartj/ehv115. Epub 2015 Apr 23. PMID 25908774

RESULTS

PARTICIPANT FLOW:
Groups:
- Home Monitoring Guided OAC: Home Monitoring is fully enabled and continuous remote surveillance data is available to investigators. Patients will be treated according to a predefined anticoagulation plan, which uses the total duration of AF/AFL combined with patients' CHADS2 score to determine the start, stop, and restart of oral anticoagulation therapy.
- Physician-Directed OAC: In Control (Group 2), Home Monitoring is active for Safety Net alerts, but the remote AF/AFL data is not revealed to the patient or treating physician. These patients receive physician-directed oral anticoagulation therapy consistent with current standards of care.
Period: Overall Study
Arm/Group | Home Monitoring Guided OAC | Physician-Directed OAC
Started | 1357 | 1361
Completed | 1006 | 1009
Not Completed | 351 | 352
Not completed — Death | 147 | 140
Not completed — Withdrawal by Subject | 152 | 139
Not completed — Lost to Follow-up | 42 | 56
Not completed — ICD device explanted | 10 | 17

BASELINE CHARACTERISTICS:
Population: All enrolled subjects
Groups:
- Total: Total of all reporting groups
Arm/Group | Home Monitoring Guided OAC | Physician-Directed OAC | Total
Number analyzed (Participants) | 1357 | 1361 | 2718
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (10.8) | 64.2 (11.5) | 64.4 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 347 | 368 | 715
  Male | 1010 | 993 | 2003

OUTCOME MEASURES:

1. Primary Outcome: Composite Primary Endpoint: Kaplan-Meier Estimate of Patients Without a Stroke, Systemic Embolism, or Major Bleed
Description: The primary endpoint is to demonstrate whether early detection of atrial arrhythmias based on BIOTRONIK Home Monitoring technology combined with a predefined anticoagulation plan in the Home Monitoring Guided OAC group is superior to the Physician-Directed OAC group reflecting conventional care and physician directed treatment of AF in terms of risk reduction of the primary composite endpoint including stroke, systemic embolism, and major bleeding events.
Time Frame: From date of enrollment until date of primary endpoint event, assessed up to study exit, with a mean treatment duration of 2.0 years
Population: Intent to treat analysis of all enrolled subjects
Measure: Number; unit: percentage of participants-Kaplan Meier
Arm/Group | Home Monitoring Guided OAC | Physician-Directed OAC
Number analyzed (Participants) | 1357 | 1361
percentage of participants-Kaplan Meier
  Kaplan-Meier estimate at 1 Year | 97.5 | 97.7
  Kaplan-Meier estimate at 2 Years | 94.8 | 95.7
  Kaplan-Meier estimate at 3 Years | 92.3 | 92.0
  Kaplan-Meier estimate at 4 Years | 90.0 | 89.4
  Kaplan-Meier estimate at 5 Years | 86.8 | 87.9
Statistical Analysis 1: Comparison: Home Monitoring Guided OAC vs Physician-Directed OAC; Test type: Superiority or Other; p = 0.732, Regression, Cox; Hazard Ratio (HR) = 1.064, 95% CI 2-sided [0.75 to 1.51]

2. Secondary Outcome: Rates of All-cause Mortality
Time Frame: Study duration from date of enrollment to date of study exit, with mean implant duration of 2.0 years
Measure: Count of Participants; unit: Participants
Arm/Group | Home Monitoring Guided OAC | Physician-Directed OAC
Number analyzed (Participants) | 1357 | 1361
Participants | 147 | 140

3. Secondary Outcome: Rate of Ischemic and Hemorrhagic Stroke
Time Frame: Study duration from date of enrollment to date of study exit, with mean implant duration of 2.0 years
Measure: Count of Participants; unit: Participants
Arm/Group | Home Monitoring Guided OAC | Physician-Directed OAC
Number analyzed (Participants) | 1357 | 1361
Participants
  Ischemic stroke | 22 | 28
  Hemorrhagic stroke | 3 | 3

4. Secondary Outcome: Rate of Fatal or Disabling and Non-disabling Stroke
Time Frame: Study duration from date of enrollment to date of study exit, with mean implant duration of 2.0 years
Measure: Count of Participants; unit: Participants
Arm/Group | Home Monitoring Guided OAC | Physician-Directed OAC
Number analyzed (Participants) | 1357 | 1361
Participants
  Fatal or disabling stroke | 9 | 11
  Non-disabling stroke | 15 | 19

5. Secondary Outcome: Rate of Major Bleeding Events
Time Frame: Study duration from date of enrollment to date of study exit, with mean implant duration of 2.0 years
Measure: Count of Participants; unit: Participants
Arm/Group | Home Monitoring Guided OAC | Physician-Directed OAC
Number analyzed (Participants) | 1357 | 1361
Participants | 46 | 34

6. Secondary Outcome: Mean Atrial Fibrillation/Atrial Flutter Burden
Time Frame: Study duration from date of enrollment to date of study exit, with mean implant duration of 2.0 years
Measure: Mean (Standard Deviation); unit: percent daily burden
Arm/Group | Home Monitoring Guided OAC | Physician-Directed OAC
Number analyzed (Participants) | 1357 | 1361
percent daily burden | 1.3 (8.2) | 1.2 (7.4)

7. Secondary Outcome: Rate of Cardioembolic and Non-cardioembolic Stroke
Time Frame: Study duration from date of enrollment to date of study exit, with mean implant duration of 2.0 years
Measure: Count of Participants; unit: Participants
Arm/Group | Home Monitoring Guided OAC | Physician-Directed OAC
Number analyzed (Participants) | 1357 | 1361
Participants
  Cardiogenic embolism | 9 | 7
  Non-cardiogenic | 5 | 8

8. Secondary Outcome: Change in Quality of Life Score
Description: Quality of Life was evaluated using the SF-36 v2 Health Survey. The SF-36 consists of eight scaled scores which correspond to the following sections: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, and mental health. Responses are recoded per a scoring key with each question having a value from 0 to 100. Scores from items in the same scale are averaged together per the scoring key to create the section and subsection (physical health and mental health) scores. For all reported scores, the lowest possible value is 0 (representing the highest disability) and the highest possible value is 100 (representing no disability). Therefore, a positive change from baseline to 1 year represents an improvement in disability, while a negative change represents a worsening of disability.
Time Frame: 1 year
Population: Subjects with paired baseline and 1 year Quality of Life scores
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Home Monitoring Guided OAC | Physician-Directed OAC
Number analyzed (Participants) | 886 | 889
Scores on a scale
  Physical health summary | 1.3 (8.8) | 0.9 (8.8)
  Mental health summary | 1.9 (11.0) | 1.6 (11.2)

9. Secondary Outcome: Mean Ventricular Heart Rate Reduction
Time Frame: 1 year
Population: Subjects with baseline and 1 year ventricular rate information
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Home Monitoring Guided OAC | Physician-Directed OAC
Number analyzed (Participants) | 877 | 878
beats per minute | 0.07 (6.31) | -0.34 (5.90)

ADVERSE EVENTS:
Time Frame: Study duration from date of enrollment to date of study exit, with a mean implant duration of 2.0 years
Description: Data for serious adverse event subcategories with an incidence of less than 1.0% are not shown. Patients could have more than one event.
Arm/Group | Home Monitoring Guided OAC | Physician-Directed OAC
Serious Adverse Events (participants affected / at risk) | 372/1357 | 374/1361
Other Adverse Events (participants affected / at risk) | 135/1357 | 139/1361
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Home Monitoring Guided OAC (N=1357) | Physician-Directed OAC (N=1361)
Congestive heart failure (Cardiac disorders) | 136 (229) | 127 (222) — With hospitalization
Arrhythmia (Cardiac disorders) | 64 (81) | 63 (77) — With hospitalization
Angina (Cardiac disorders) | 42 (60) | 53 (65) — With hospitalization
Dyspnea (Cardiac disorders) | 17 (20) | 26 (26) — With hospitalization
Coronary artery disease (Cardiac disorders) | 28 (31) | 18 (21) — With hospitalization
Myocardial infaction (Cardiac disorders) | 26 (30) | 35 (39) — With hospitalization
Cardiac arrest (Cardiac disorders) | 23 (24) | 27 (27) — With hospitalization or resulting in death
Stroke (Nervous system disorders) | 22 (25) | 30 (31) — With hospitalization, resulting in death, or persistent/significant disability
Gastrointestianal bleeding (Vascular disorders) | 23 (25) | 18 (19) — With hospitalization or results in death
Upgrade to CRT-D device (Surgical and medical procedures) | 25 (26) | 18 (18) — With hospitalization
Device replacement (Surgical and medical procedures) | 15 (15) | 9 (9) — With hospitalization
Lead replacement or repositioning (Surgical and medical procedures) | 16 (17) | 11 (12) — With hospitalization
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Home Monitoring Guided OAC (N=1357) | Physician-Directed OAC (N=1361)
Congestive Heart Failure (Cardiac disorders) | 22 (39) | 25 (51) — Not requiring hospitalization
Arrhythmia (Cardiac disorders) | 52 (84) | 53 (74) — Not requiring hospitalization
Angina (Cardiac disorders) | 32 (49) | 34 (48) — Not requiring hospitalization
Dyspnea (Cardiac disorders) | 19 (19) | 18 (19) — Not requiring hospitalization
Device replacement (Surgical and medical procedures) | 29 (29) | 35 (35) — Done as an outpatient procedure (not requiring hospitalization)

LIMITATIONS AND CAVEATS:
Study stopped early when primary endpoint met futility criteria. Continuation may have changed the outcome; however, unlikely to demonstrate a meaningful clinical benefit. Interpretation of secondary endpoints should be approached with caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No